CLINICAL TRIAL: NCT04697407
Title: BREGS - IL-2 Signaling and Polarization of Regulatory LBs: Involvement in Multiple Sclerosis
Brief Title: IL-2 Signaling and Polarization of Regulatory LBs: Involvement in Multiple Sclerosis
Acronym: BREGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 35RC20_9867_BREGS
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MS Patients (Experimental): Patients with MS at any stage and for any type of MS : MS at the onset of the disease, Clinically isolated syndrome (CIS), Relapsing-remitting MS (RRMS), Primary progressive MS (PPMS), Secondary progressive MS (SPMS)
  Interventions: Biological: Blood sampling; Biological: CSF sampling
- non MS Patients (Active Comparator): Patients with a neurological and immunological disease except MS.
  Interventions: Biological: Blood sampling; Biological: CSF sampling
- Healthy volunteers (Active Comparator)
  Interventions: Biological: Blood sampling

INTERVENTIONS:
Biological: Blood sampling — In all groups, 80 ml of blood will be collected. For patients, this will be done during routine cares.
Biological: CSF sampling — Only in both patients groups whom will have a CSF sampling in routine care, some CSF will be collected for the study in addition, with a limit of 5 ml for routine care and study.
  Arms: MS Patients; non MS Patients

SUMMARY:
Multiple sclerosis (MS) has long been considered a disease mediated primarily by CD4+ T cells. However, recent clinical trials demonstrating significant efficacy of B-lymphocyte depletive therapies have highlighted the major role of this cell population in the development of MS. Among B-Ls, regulatory ("anti-inflammatory") B-Ls (Bregs) have protective functions in autoimmune diseases including MS, however the mechanisms that regulate the development and function of Bregs are poorly characterized. In our research laboratory (INSERM UMR1236), one of the lines of research focuses on the role of interleukin-2 (IL-2) signaling in the fate of the B lymphocyte. Numerous studies conducted in both human and mouse models of MS demonstrate the major role of this IL-2/IL2R signaling pathway in the pathogenesis of autoimmune diseases.

The hypothesis is that IL-2/IL2R pathway could contribute, by a mechanism intrinsic to B lymphocytes, to the development of autoimmune diseases such as MS.

While a defect in IL-2 signaling plays a critical role in the pathogenesis of MS, the impact of this defective signaling on regulatory B lymphocyte populations, which has been shown to play a protective role in the development of the disease, has never been studied. This study could help establish a new mechanism predisposing patients to develop the disease.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is an autoimmune disease of the central nervous system (CNS) that is the leading cause of non-traumatic disability in young adults. Pathophysiopathologically, MS has long been considered a disease mediated primarily by CD4+ T cells. However, recent clinical trials demonstrating significant efficacy of B-lymphocyte (B-lymphocyte) depletive therapies have highlighted the major role of this cell population in the development of MS. Thus, it has been shown that these cells, in addition to their ability to secrete pathogenic antibodies, produce pro-inflammatory cytokines in this disease, and an imbalance between these potentially pathogenic pro-inflammatory B-Ls and regulatory ("anti-inflammatory") B-Ls (Bregs) has been suggested.

Bregs have protective functions in autoimmune diseases including MS, however the mechanisms that regulate the development and function of Bregs are poorly characterized. In our research laboratory (INSERM UMR1236), one of the lines of research focuses on the role of interleukin-2 (IL-2) signaling in the fate of the B lymphocyte. Our team has thus demonstrated that this cytokine, essentially produced by CD4+ T lymphocytes, triggers the differentiation of naïve human B cells in vitro into plasma cells. And, more recently, the analysis of the early response of BLs in mice disabled for the IL-2 receptor specifically in mature BLs (Il2rbfl/flCD19cre/+) suggests a role of IL-2 in the acquisition of suppressive/regulatory functions. In addition, numerous studies conducted in both human and mouse models of MS demonstrate the major role of this IL-2/IL2R signaling pathway in the pathogenesis of autoimmune diseases.

The hypothesis is that IL-2 signaling induces the polarization and/or regulatory function of Bregs in vivo and that deregulation of this IL-2/IL2R pathway could contribute, by a mechanism intrinsic to B lymphocytes, to the development of autoimmune diseases such as MS.

While a defect in IL-2 signaling plays a critical role in the pathogenesis of MS, the impact of this defective signaling on regulatory B lymphocyte populations, which has been shown to play a protective role in the development of the disease, has never been studied. This study could help establish a new mechanism predisposing patients to develop the disease.

The objective of this study is the analysis of the Bregs population in the blood of MS patients (at the diagnostic stage and in different forms) who are untreated compared to controls who are healthy in various aspects.

ELIGIBILITY:
About the patients,Inclusion Criteria :

* Patients at the onset of illness :
* With a strong suspicion of MS requiring an LP to confirm the diagnosis (suggestive neurological symptoms AND more than two typical lesions on MRI) ; OR
* MS patients (untreated RR, SP or PP) :
* With MS that meets the MacDonald 2017 criteria;
* With relapsing-remitting (RR), secondary-progressive (SP) or primary-progressive (PP) MS; OR
* Non-MS patients :
* Presenting a non MS neurological inflammatory disease (meningitis, neurolupus, neurosarcoidosis, autoimmune encephalitis, acute polyradiculoneuritis);
* Benefiting from an LP for diagnostic or monitoring purposes;

AND

* At least 18 years old;
* Without immunomodulating or immunosuppressive background treatment for at least 3 months;
* Without systemic corticosteroid treatment for at least 3 months;
* Having signed a free, informed and written consent.
* Affiliated with a social security system

About healthy volunteers, inclusion criteria :

* At least 18 years old;
* Having signed a free, informed and written consent.
* Affiliated with a social security system

Exclusion Criteria:

For all groups

* Pregnancy ;
* Breastfeeding ;
* Persons of full age subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.

Healthy volunteers :

* Absence of autoimmune pathologies
* Without immunomodulating or immunosuppressive background treatment for at least 3 months;
* Without systemic corticosteroid treatment for at least 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Frequency of Bregs in blood of MS patients | 1 month
  Comparison of the frequency of Bregs in the blood of untreated MS patients (at the diagnostic stage and in different forms of MS: Relapsing-remitting (RR), Primary Progressive (PP) and Secondary Progressive (SP)) compared to healthy controls matched for age and gender.

SECONDARY OUTCOMES:
Frequency of Bregs in the CSF of MS patients | 1 month
  Comparison of the frequency of Bregs in the CSF of early MS patients to the frequency of Bregs in the CSF of patients with other non-MS inflammatory neurological diseases.
Comparison of IL-2, soluble IL2RA, IL-10, IL-21 and IL-5 protein concentrations | 1 month
  Comparison of IL-2, soluble IL2RA, IL-10, IL-21 and IL-5 protein concentrations in blood and/or CSF of MS patients to protein concentration of patients with inflammatory neurological non MS disease and to protein concentration in blood of healthy volunteers
Comparison of the concentrations in Igs | 1 month
  Comparison of the concentrations in immunoglobulins in blood and/or CSF of MS patients to protein concentration of patients with inflammatory neurological non MS disease and to immunoglobulin concentration in blood of healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Laure Michel, Md, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No